CLINICAL TRIAL: NCT01888458
Title: Antifungal Prophylaxis With Micafungin After Cord Blood Allogeneic Stem Cell Transplantation
Brief Title: Antifungal Prophylaxis With Micafungin After Cord Blood Allogeneic Stem Cell Transplantation (MycaCOORD)
Acronym: MycaCOORD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC13_0008
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Invasive Fungal Infection
Keywords: Adult; allo-Stem Cell Transplantation; Cord Blood
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Micafungine (Experimental)
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — All patients meeting selection criteria will receive micafungin IV. Prophylaxis will start within 48 hours of the beginning of the transplant-related conditioning regimen until 5 days after recovery from neutropenia (ANC ≥ 500/µl), or occurrence of an IFI, or up to 42 days, or withdrawal for any reason (e.g. patient's or investigator's decision, development of intolerance, death), whichever come first

SUMMARY:
Infections due to post transplant immune deficiency are a major problem following allogeneic stem cell transplantation (Allo-SCT), particularly in patients receiving cord blood transplant (CB). Duration of neutropenia is one of the most important risk factor for invasive fungal infection (IFI). In this setting, Micafungin has been approved for antifungal prophylaxis for patients undergoing Allo-SCT. In a randomized, double-blind, comparative, phase III trial, the overall efficacy of micafungin was superior to that of fluconazole as antifungal prophylaxis during the neutropenic phase after Allo-SCT. However, very few patients in this study received a CB transplant.

This is phase IIb, prospective, open-label, non-comparative study to assess the safety of micafungin when use in prevention of IFI in neutropenic patients receiving allo-SCT using CB as source of stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients receiving allo-Stem Cell Transplantation using Cord Blood as source of stem cells (cf conditioning regimen recommendation).
* Sex male or female
* Age between 18 and 65 years at the time of signing the informed consent form.
* Diagnosis of an hematologic disease for who a allograft decision has been taken
* not having a (HLA)-matched related or unrelated donor within two month after complete remission achievement
* Able to understand and voluntarily sign an informed consent form.
* Subjects affiliated with an appropriate social security system
* Male, female without childbearing potential or negative urine pregnancy test at the screening visit prior to beginning the treatment. Women of childbearing potential must be following adequate contraceptive measures. Men must agree to use an acceptable method of contraception (for themselves or female partners) for the duration of the study
* Each subject will weigh 40 kg or more

Exclusion Criteria:

* Any suspected or documented invasive fungal infection at study entry or at any time prior to study entry
* Use of any systemic antifungal therapy within 72 hours prior to study entry
* Known history of allergy, hypersensitivity or intolerance to echinocandin agents
* Patient with any medical, psychological or social condition, which in the opinion of the investigator could increase the risk to the patient, or decrease the chance of obtaining satisfactory data to achieve the objectives of this study.
* Participation in a study testing a new drug or a new conditioning
* HIV, HBV or HCV positive
* Pregnant or breast feeding females.
* Subject protected by law.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety | 50 days
  Safety assessed by the incidence and type of adverse events (AE) occurring during the course of prophylaxis treatment, AE related to study drug, AE leading to study drug discontinuation, and evolution of vital signs and biological parameters.

SECONDARY OUTCOMES:
Incidence of Invasive Fungal Infection | 50 days
  Incidence of Invasive Fungal Infection (IFI) at the end of prophylaxis period and at the end of the 4-week follow-up period
Incidence of fever of unknown origin | 50 days
  Incidence of fever of unknown origin requiring empirical antifungal treatment during prophylaxis period
Survival rate | 50 days
  Survival rate and incidence of mortality related to IFI from the start of prophylaxis until the end of the 4-week follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricette MICHALLET, PU PH, Principal Investigator — Hospices Civils de Lyon; Sabine FURST, PH, Principal Investigator — Institut Paoli et Calmette (Marseille); Valérie COITEUX, PU PH, Principal Investigator — CHRU de Lille; Stéphane VIGOUROUX, PH, Principal Investigator — University Hospital, Bordeaux; Mohamad MOHTY, PU PH, Principal Investigator — AP-HP Saint Antoine; Thomas GASTINNE, PH, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France